CLINICAL TRIAL: NCT05434494
Title: The Effect of Remifentanil on ED95 of Remimazolam for Loss of Consciousness in Adult Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AJIRB-MED-INT-22-008
Record Dates: First submitted 2022-06-20; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Remimazolam
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remifentanil group (Active Comparator): Start the continuous infusion of 25cc of remifantanil (labeled as a test drug) by TCI mode ( the target effect site concentration is 2.0).
  While slowly injecting the prescribed dose of remimazolam over 30 seconds, observe whether it responds to the investigator's oral commands and the disappearance of the eyelash reflex for 3 minutes after administering the drug. Success in inducing loss of consciousness during anesthesia is defined as the loss of both verbal command response and eyelash reflex within 3 minutes after infusion, otherwise it is considered a failure.
  The dose of remimazolam is initially 0.15 mg/kg and the next experimental dose is determined according to the biased coin design up-and-down sequential method. The standard deviation of this study is 0.05 mg.
  Interventions: Drug: Remimazolam; Drug: remifantanil
- control group (Placebo Comparator): Start the continuous infusion of 25cc of normal saline (labeled as a test drug).
  While slowly injecting the prescribed dose of remimazolam over 30 seconds, observe whether it responds to the investigator's oral commands and the disappearance of the eyelash reflex for 3 minutes after administering the drug. Success in inducing loss of consciousness during anesthesia is defined as the loss of both verbal command response and eyelash reflex within 3 minutes after infusion, otherwise it is considered a failure.
  The dose of remimazolam is initially 0.15 mg/kg and the next experimental dose is determined according to the biased coin design up-and-down sequential method. The standard deviation of this study is 0.05 mg.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is injected for 30 seconds and the experimental dose will be determined according to the biased coin design up-and-down sequential method.
  If loss of consciousness is successful, the dose of the next intravenous dose of the next study subject will be reduced from the previous dose with a probability of 1/19 or the same as the previous dose with a probability of 18/19.
Drug: remifantanil — 25cc infusion drug will be prepared (labeled as test drug) and infused with TCI mode. The target effect site concentration is 2.0 ng/ml.
  Arms: remifentanil group

SUMMARY:
This study prospectively uses the biased coin technique to investigate the effect of concomitant administration of remifentanil on the 95% effective dose of intravenous remimazolam (Effective dose 95 [ED95]) required for loss of consciousness during anesthesia induction. .

ELIGIBILITY:
Inclusion Criteria:

* The adult patients who are scheduled to surgery under general anesthesia

Exclusion Criteria:

* Severe obesity (BMI > 30 kg/m2)
* Allergy to remimazolam or remifentanil
* Under conditions which make it difficult to respond to the investigator's verbal commends like hearing impairment, etc.
* Patients with general conditions are more than ASA class III
* Patients with brain disease (dementia, cerebral infarction, etc.)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Remimazolam dose at which loss of consciousness occurs | 3 min after remimazolam injection
  While slowly injecting the prescribed dose of remimazolam over 30 seconds, observe whether it responds to the investigator's oral commands and the disappearance of the eyelash reflex for 3 minutes after administering the drug. Success in inducing loss of consciousness during anesthesia is defined as the loss of both verbal command response and eyelash reflex within 3 minutes after infusion, otherwise it is considered a failure.

SECONDARY OUTCOMES:
Time to loss of consciousness | time after injection of remimazolam to loss of conciousness
  After injection of remimazolam, the investigator concludes the successful loss of consciousness (not respond to oral commands and the disappearance of the eyelash reflex); From remimazolam injection until loss of consciousness occurs